CLINICAL TRIAL: NCT00239551
Title: Effect of Prevacid on Prostaglandin Levels in the Gastric Mucosa of Patients With Stress Ulcer
Brief Title: Effect of Prevacid on Prostaglandin Levels in Patient With Stress Ulcer
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: TAP Pharmaceutical Products Inc. (Industry)
Responsible Party: Principal Investigator, Dr. Qiang Cai MD/PhD, Professor, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 623-2005
Record Dates: First submitted 2005-10-13; First posted 2005-10-17 (Estimated); Last update posted 2013-07-31 (Estimated); Status verified 2013-07

CONDITIONS: Stomach Ulcer
Keywords: gastric stress ulcer; Prevacid; Prostaglandin
MeSH Terms: conditions — Stomach Ulcer; Duodenal Ulcer | interventions — Lansoprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Prevacid (Experimental): Effect of Prevacid at 8 weeks; EGD(esophagogastroduodenal endoscopy) at day 1 & EGD at 8 weeks
  Interventions: Drug: Prevacid

INTERVENTIONS:
Drug: Prevacid — Effect of Prevacid on prostaglandin levels at 8 weeks; EGD (esophagogastroduodenal endoscopy) with biopsy at day 1 & EGD with biopsy at 8 weeks
  Other Names: Lansoprazole

SUMMARY:
The purpose of this study is to measure the prostaglandin levels in patients with stress ulcer and the effect of Prevacid on prostaglandin levels in patients with stress ulcer.

DETAILED DESCRIPTION:
The prostaglandin system plays an important role in the gastric mucosa to strengthen its resistance against injury. Critically ill patients are at greatest risk of developing stress-related gastric mucosal lesions. Although the levels of prostaglandins in gastric mucosa in patients with stressed animal has been studied, prostaglandin levels in the gastric mucosa in patients with stress ulcer have not been studied and the effect of Prevacid on prostaglandin levels in gastric mucosa from patients with stress ulcer is unknown.

We hypothesize that prostaglandin levels are low in the gastric mucosa in patients with stress ulcer, and Prevacid is an effective agents in increasing prostaglandin levels in the gastric mucosa in stress stress ulcer.

Comparison(s): The prostaglandin levels in patients who treated with Prevacid for stress ulcer, compared to the prostaglandin levels in patients who treated with H2 blocker for stress ulcer.

ELIGIBILITY:
Inclusion Criteria:

* Patients in ICU with documented gastric stress ulcer by endoscopic examination, including patients with H. Pylori infection;
* Patients have no known ulcer within 8 weeks prior to be admitted to ICU;
* Patients not on any PPI for 4 weeks prior to the study;
* Patients or family be consented for the study.

Exclusion Criteria:

* Patients have gastric ulcer within 8 weeks prior to be admitted to ICU;
* Patients have gastric cancer confirmed by pathology;
* Patients on one of the PPIs already;
* Patients on any of the Non-steroidal Antiinflammatory Drugs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2005-10; Primary Completion 2006-10 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
the effect of Prevacid on prostaglandin levels at 8 weeks | 8 weeks

SECONDARY OUTCOMES:
esophagogastroduodenal endoscopy(EGD) with biopsy at day 1; EGD with biopsy at 8 weeks | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Qiang Cai, MD, PhD, Principal Investigator — Emory University; Vincent W Yang, MD, PhD, Study Director — Emory University
Locations (1):
- Emory University School of Medicine, Atlanta, Georgia, United States